CLINICAL TRIAL: NCT01001793
Title: Evaluation of the Levacor™ Ventricular Assist Device as a Bridge to Cardiac Transplantation
Brief Title: Levacor™ Ventricular Assist Device (VAD) Bridge to Transplant Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Commercial considerations relating to required device modifications.
Sponsor: World Heart Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEV01
Record Dates: First submitted 2009-10-24; First posted 2009-10-27 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-09

CONDITIONS: Refractory Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Levacor Ventricular Assist Device — Surgical procedure

SUMMARY:
The Levacor™ Ventricular Assist Device (VAD) has been designed for mechanical circulatory support in heart failure patients. The purpose of this clinical study is to determine its safety and efficacy as a bridge to transplant (BTT) in cardiac transplant candidates with presumed non-reversible left ventricular failure.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least 18 years of age at the time of VAD implantation.
2. Listed for cardiac transplantation as UNOS Status 1A or 1B at the time of VAD implantation or within 72 hours of VAD implantation.
3. Body Surface Area (BSA) 1.2 m2 or greater.
4. If female of childbearing potential must have negative pregnancy test.
5. Patient has signed an Informed Consent.

Exclusion Criteria:

1. Unacceptable surgical risk according to Principal Investigator.
2. Intolerance or contraindication to anticoagulation or antiplatelet therapies.
3. Excessive risk of bleeding as evidenced by INR > 2.3, or PTT > 45 sec, or platelet count < 50,000 U, unresponsive to treatment.
4. Excessive neurologic risk documented as TIA within the last 3 months or stroke within the last 6 months.
5. Evidence of any of the following indicators of end-organ dysfunction: total bilirubin > 4 mg/dL, ALT/AST > 3 times upper limit normal, serum creatinine >3.5 mg/dL.
6. Fixed pulmonary hypertension with a most recent PVR > 5 Wood units unresponsive to pharmacological intervention.
7. Severe chronic obstructive pulmonary disease as evidenced by an FEV1 < 1.0 L or restrictive lung disease or prolonged (> 48 hours) intubation.
8. Presence of mechanical aortic valve that will not be converted to a bioprosthesis during VAD implantation.
9. Planned concomitant surgical procedures other than aortic valve repair or tissue valve placement to treat moderate to severe aortic insufficiency, tricuspid valve repair, mitral valve repair, critical lesion CABG, LV thrombectomy (apical), closure of persistent foramen ovale, atrial septal defect.
10. Cardiogenic shock secondary to acute myocardial infarction.
11. Presence of ongoing mechanical circulatory support other than intra-aortic balloon counterpulsation.
12. Presence of uncontrolled infection.
13. BMI > 40 kg/m2.
14. Significant peripheral vascular disease accompanied by pain at rest, extremity ulceration or disabling claudication.
15. Illness, other than heart disease, that would limit survival to less than 1 year.
16. Pulmonary embolus < 2 weeks before VAD implant.
17. Poor/compromising nutritional status in judgment of Principal Investigator.
18. Participation in another clinical trial that, according to the Principal Investigator, is likely to affect the Study outcome or confound the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Success is defined as any one of the following: survival to cardiac transplantation prior to 180 days, survival on device to 180 days, device removal for recovery and survival to 60 days after device removal | 6 months

SECONDARY OUTCOMES:
Survival to transplant | 6 months
Survival 30 days post-transplant | 6 months
Survival while on device | 6 months
Incidence of adverse events while on device | 6 months
Device reliability | 6 months
Reoperations | 6 months
Functional status | 6 months
Quality of life | 6 months
Neurocognitive evaluation | 6 months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Tampa General Hospital, Tampa, Florida
  - Jewish Hospital, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - University of Utah Hospital, Salt Lake City, Utah
  - Inova Fairfax Hospital/Inova Heart & Vascular Institute, Falls Church, Virginia